CLINICAL TRIAL: NCT06798324
Title: Using Non-Invasive Brain Stimulation (tDCS) as an Adjunct to Varenicline for the Treatment of Tobacco Dependence: a Randomized Controlled Trial
Brief Title: tDCS Plus Varenicline for Smoking Cessation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Laurie Zawertailo, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 081-2024; 508405 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-01-08; First posted 2025-01-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Nicotine Dependence; Tobacco Smoking; Smoking Cessation; Nicotine Use Disorder; Tobacco Use Disorder; Substance Use Disorders
Keywords: Smoking; Tobacco Use Disorder; Smoking Cessation; Substance Use Disorders; Brain Stimulation; Transcranial Direct Current Stimulation; Tobacco Cigarettes; tDCS; Varenicline
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking; Smoking Cessation; Substance-Related Disorders; Smoking | interventions — Varenicline; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental Group (Active tDCS plus Varenicline) (Active Comparator): The experimental group will receive active tDCS sessions plus 12 weeks of 1 mg varenicline bid. Participants will start varenicline treatment on the same day as the first tDCS session, and will follow a standard dose escalation schedule. The tDCS treatment schedule includes 10 daily sessions for the first 2 weeks (M to F), followed by 5 single bi-weekly booster sessions for the remainder of the treatment period. Participants will come in-person for two follow-up sessions to assess smoking behaviour at 6- and 12-months post-treatment.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS); Drug: Varenicline 1mg BID
- Control Group (Sham Comparator): The control group will receive sham (fake) tDCS sessions plus 12 weeks of 1 mg varenicline bid. Participants will start varenicline treatment on the same day as the first tDCS session, and will follow a standard dose escalation schedule. The tDCS treatment schedule includes 10 daily sessions for the first 2 weeks (M to F), followed by 5 single bi-weekly booster sessions for the remainder of the treatment period. Participants will come in-person for two follow-up sessions to assess smoking behaviour at 6- and 12-months post-treatment.
  Interventions: Drug: Varenicline 1mg BID; Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation. Active tDCS involves brief (e.g., 20-min) application of weak electric current (e.g., 2 mA) to the scalp. The tDCS device that will be used for this study is the Soterix 1x1 mini-CT.
  Arms: Experimental Group (Active tDCS plus Varenicline)
Drug: Varenicline 1mg BID — Varenicline is the most effective approved treatment for quitting smoking. Varenicline as per standard prescribing for dose escalation (i.e. Days 1 to 3: 0.5 mg once daily; Days 4 to 7: 0.5 mg twice daily; Days 8 to end of treatment: 1 mg twice daily) will be given concurrently over the same 2 weeks as the tDCS protocol and continue for an additional 10 weeks as per standard treatment duration recommended on the product monograph for a total of 12 weeks of varenicline treatment. Dose adjustments due to adverse events will be allowed (i.e. decrease to 0.5 mg twice daily).
  The target quit date for smoking cessation will be on the last day of the two weeks of daily tDCS which corresponds to the recommended quit date after starting varenicline treatment.
  Other Names: Champix; Chantix
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Sham tDCS consists of 30s of 2 mA at the beginning and at the end of the 6 session (ramp up and down), then receiving 0 mA stimulation for the middle 19 min. The tDCS device that will be used for this study is the Soterix 1x1 mini-CT.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to determine if active transcranial direct current stimulation (tDCS) plus varenicline is an effective, safe and accessible treatment option for smoking cessation. The main questions this trial aims to answer are:

1. Does active tDCS plus varenicline improve short-term and long-term smoking abstinence rates compared to sham tDCS plus varenicline?
2. Are the safety profiles between active tDCS plus varenicline and sham tDCS plus varenicline different?

The tDCS treatment schedule includes 10 daily sessions for the first 2 weeks (M to F), followed by 5 single bi-weekly booster sessions for the remainder of the treatment period. Participants will come in-person for two follow-up sessions to assess smoking behaviour at 6- and 12-months post-treatment.

DETAILED DESCRIPTION:
Smoking remains the leading cause of lung cancer globally, with cigarette smokers being about 20 times more likely to develop lung cancer than non-smokers. Despite the availability of effective treatments and extensive public health efforts, quitting smoking remains a significant challenge. Varenicline is currently the most effective medication for smoking cessation, yet most users relapse within the first year. No new medications for smoking cessation have come to market in the past two decades, and as such there is a critical need to optimize existing treatments. Combining treatment modalities can produce therapeutic synergism and improve overall treatment outcomes. Non-invasive brain stimulation techniques have become a popular area of research as a treatment option for substance use disorders with growing evidence of their effectiveness for a variety of addictions. One of these techniques, transcranial direct current stimulation (tDCS), has demonstrated potential in modulating the neuroadaptations associated with chronic smoking and relapse risk. A prior pilot study in our lab found that adjunct active tDCS doubled varenicline's effectiveness at end of treatment. Therefore, the objectives for this trial are as follows:

1. To determine the short-term efficacy of active anodal tDCS to the left DLPFC plus varenicline compared to sham tDCS plus varenicline.
2. To determine the effect of active anodal tDCS to the left DLPFC plus varenicline on sustained abstinence over time.
3. To determine the safety of active anodal tDCS to the left DLPFC plus varenicline compared to sham tDCS plus varenicline.

This study will be a double-blind sham-controlled randomized clinical trial whereby 160 daily cigarette smokers will be recruited. After confirming eligibility at an assessment visit, participants will be randomized (1:1) to one of two groups: 1) Experimental group of active tDCS sessions plus 12 weeks of 1 mg varenicline bid (n=80); and 2) Control group of sham tDCS sessions plus 12 weeks of 1 mg varenicline bid (n=80). Participants will start varenicline treatment on the same day as the first tDCS session, and will follow a standard dose escalation schedule. The tDCS treatment schedule includes 10 daily sessions for the first 2 weeks (M to F), followed by 5 in-person bi-weekly booster sessions for the remainder of the treatment period, and then 2 in-person follow-up sessions to assess smoking behaviour at 6- and 12-months post-treatment. At the 1st daily session, participants will come in-person to be trained on using the tDCS device and provided with a study kit including all relevant study equipment. The following 8 daily sessions will occur remotely, and be monitored by research personnel over Webex. The 10th daily tDCS session will occur in-person, with participants returning the study kit. All 5 bi-weekly booster sessions will occur in-person. Total Study duration (with follow-up) is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide informed written consent
* Stated willingness to comply with all study procedures
* Age 18-85 years
* Smoke ≥ 8 cigarettes per day (CPD)
* Is seeking treatment for tobacco dependence
* Willing to attend the required clinic appointments (Two consecutive weeks, Monday through Friday)
* Otherwise healthy (i.e. not suffering from any major illness/condition that would impact their participation in the study)

Exclusion Criteria:

* Use of smoking cessation medication (e.g. buproprion, varenicline, NRT, cytisine) in the past 3 months
* Current regular use of nicotine-containing products besides cigarettes (e.g. electronic cigarettes, etc.)
* Unstable psychiatric illness that would adversely impact study participation and compliance (determined by the QI)
* History of seizures/epilepsy
* Lifetime history of concussions or head traumas
* Current pregnancy or plans to become pregnant
* Current pacemakers or implanted electrical devices
* Current metal embedded in the skull
* Presence of skin lesions, open wounds, or bruising at stimulation sites; or
* Contraindications to varenicline use (e.g. pregnant/breastfeeding, alcohol dependence, kidney disease/renal impairment, known hypersensitivity to varenicline)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2028-01-20 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
30-Day Continuous Abstinence at End-Of-Treatment | Week 9-12
  Proportion of the sample that has been abstinent from smoking for 30 days at end of treatment (treatment weeks 9-12), verified with a negative urinary cotinine test.

SECONDARY OUTCOMES:
Long-term Sustained Abstinence at Follow-Up | Weeks 9-26 and Weeks 9-52
  Continuous abstinence at 6-months (weeks 9 to 26) and 12-month (weeks 9 to 52) follow-up (verified with a negative urinary cotinine test).
Adverse events | Week 1-52
  Adverse events will be recorded throughout the treatment and in follow-up visits.
Working Memory Scores | Week 1-52
  The N-back Task will be used throughout the study to evaluate changes in working memory.
Attentional Bias | Week 1-52
  Attentional bias towards smoking cues, sensation-seeking cues, and negative affect cues will be evaluated throughout the study using eye-tracking technology.
Inhibitory Control Scores | Week 1-52
  Inhibitory control will be evaluated throughout the study using the Stop Signal Task and the Sustained Attention to Response Task.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Zawertailo, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zawertailo L, Zhang H, Rahmani N, Rajji TK, Selby P. Active versus sham transcranial direct current stimulation (tDCS) as an adjunct to varenicline treatment for smoking cessation: Study protocol for a double-blind single dummy randomized controlled trial. PLoS One. 2022 Dec 8;17(12):e0277408. doi: 10.1371/journal.pone.0277408. eCollection 2022. PMID 36480510
- [Background] Zhang H, Rajji TK, Selby P, Melamed O, Attwells S, Zawertailo L. Augmenting varenicline treatment with transcranial direct current stimulation (tDCS) increases smoking abstinence rates at end of treatment. Brain Stimul. 2023 Jul-Aug;16(4):1083-1085. doi: 10.1016/j.brs.2023.07.001. Epub 2023 Jul 3. No abstract available. PMID 37406928